CLINICAL TRIAL: NCT00510705
Title: Chronic Inflammatory Activation in Fat Tissue: An Atherogenic Factor in Severe Coronary Artery Disease
Acronym: KFO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Axel Linke, Co-Investigator, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0816-2007
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2014-12

CONDITIONS: Severe Coronary Artery Disease; Obesity; Impaired Glucose Tolerance
Keywords: adiposity
MeSH Terms: conditions — Coronary Artery Disease; Obesity; Glucose Intolerance | interventions — Exercise; Metformin; Thiazolidinediones

ARMS (4):
- 1 (Other): Regular physical exercise training alone
  Interventions: Other: exercise training
- 2 (Other): Regular physical exercise training + metformin
  Interventions: Other: exercise training + metformin
- 3 (Other): Regular physical exercise training + glitazone
  Interventions: Other: exercise training + glitazone
- 4 (No Intervention): Control

INTERVENTIONS:
Other: exercise training — physical exercise training on a bicycle ergometer daily for 4 weeks
  Arms: 1
Other: exercise training + metformin — physical exercise training on a bicycle ergometer + metformin (2 x 850 mg) daily for 4 weeks
  Arms: 2
Other: exercise training + glitazone — physical exercise training on a bicycle ergometer + glitazone daily for 4 weeks
  Arms: 3

SUMMARY:
Chronic inflammatory activation in fat tissue can be the link between adiposity and an increased risk for atherosclerosis. The aim of this study is to investigate how molecular alterations in fat tissue can be influenced by regular physical exercise training alone or in combination with a medical therapy (glitazone or metformin) in obese patients with severe coronary artery disease (CAD) and impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Either impaired glucose tolerance (2 hour plasma glucose concentration > 7.8 and < 11.1 mmol/L during an oral glucose tolerance test) or impaired fasting plasma glucose concentration ( > 6.0 and < 7.0 mmol/L)
* Body mass index (BMI) > 25
* Severe coronary artery disease determined by coronary angiography
* Male patients aged 35-75 years

Exclusion Criteria:

* Diabetes mellitus type I
* Diabetes mellitus type II in combination with glycosylates hemoglobin > 6.0%, previous medication with oral antidiabetic agents or insulin, fasting plasma glucose concentration > 11.0 mmol/L
* Unstable angina pectoris
* Myocardial infarction within the last 4 weeks
* Reduced left-ventricular systolic function < 30%

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
change in endothelial function in severe coronary artery disease | 4 weeks

SECONDARY OUTCOMES:
change in metabolic parameters | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schuler, Prof. of Medicine, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany